CLINICAL TRIAL: NCT04724798
Title: Population Pharmacokinetics of Tigecycline in Patients Treated With ECMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Zhenhua Zen, Associate Professor, Nanfang Hospital, Southern Medical University
Other Study IDs: NFEC-2020-021
Record Dates: First submitted 2021-01-19; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Extracorporeal Membrane Oxygenation; Pharmacokinetics; Tigecycline

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tigecycline is a commonly used antibiotic in critically ill patients. The pharmacokinetics (PK) of tigecycline in intensive care unit (ICU) patients can be affected by severe pathophysiological changes so that standard dosing might not be adequate. At present, a number of studies have reported that ECMO will affect the PK of anti-infective drugs and lead to treatment failure. The purpose of this study was to describe the population PK of tigecycline in patients treated with ECMO and to evaluate the relationship between individual PK parameters and patient covariates.

ELIGIBILITY:
Inclusion Criteria:

* critically ill hospitalized males or nonpregnant females aged ≥18 years with severe infections which the treating clinician was treating with tigecycline.

Exclusion Criteria:

* People who had taken tigecycline in the past week
* People who were pregnant
* People who had coagulation dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill hospitalized males or nonpregnant females aged ≥18 years with severe infections which the treating clinician was treating with tigecycline.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Serum drug concentration of tigecycline | predose, 2 min, 5 min, 15 min, 30 min, 1 hour, 3 hours, 6 hours, 12 hours, and 24 hours post-dose
  Serum drug concentration at different time points in each adult ICU patient treated with ECMO

CONTACTS AND LOCATIONS:
Locations (1):
- Southern medical university Nanfang hospital, Guangzhou, China